CLINICAL TRIAL: NCT02256449
Title: Registry of Patients With Bioresorbable Device in Daily Clinical Practice. REPARA Study
Brief Title: REPARA Study: REgistry of PAtients With bioResorbable Device in Daily Clinical prActice
Acronym: REPARA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sección Hemodinamica y Cardiologia Intervencionista (Other)
Responsible Party: Sponsor
Other Study IDs: COR-BVS-2013-01
Record Dates: First submitted 2014-09-23; First posted 2014-10-03 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Coronary Artery Lesions With Implantation of Coronary Device
Keywords: Coronary artery disease; angioplasty; bioresorbable device
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- BVS patients: Use of bioresorbable coronary device, according to the indications of use, in daily clinical practice, in patients undergoing PCI in de novo coronary artery lesions.

SUMMARY:
A multicentre, observational, prospective device registry, with no control group, designed to evaluate the efficacy and safety of the bioresorbable coronary device, used according to the indications of use, in daily clinical practice in a consecutive number of patients undergoing PCI in de novo coronary artery lesions. A total of 1,500 patients are planned to be included in the registry.

DETAILED DESCRIPTION:
The patients will be included consecutively at each site for one year. They will be individuals from both sexes, requiring endovascular intervention and meeting the authorised criteria for the indications of use of the device to be used and where dual anti-platelet therapy (DAPT) with aspirin and thienopyridines is considered.

STUDY OBJECTIVES To evaluate the MACE rate after implantation of the bioresorbable coronary device in patients with de novo coronary artery lesions, where a follow-up of 12 months will be performed.

Primary objective:

MACE rate at 12 months of follow-up:

Cardiac death Myocardial infarction TLR driven by ischaemia of the lesion treated or of the region of 5 mm proximally or distally to the site of implantation of the device (ID-TLR).

Secondary objectives:

* Angina
* Death due to any cause.
* Myocardial infarction of any type (MI: QMI, NQMI, TV, NTV)
* All TLR driven or not by ischaemia
* All TVR driven or not by ischaemia.
* All coronary revascularisations performed (PCI vs CABG)
* Device thrombosis (acute, sub-acute, late) and evidence (definitive, probable, possible).
* Immediate success of the device.
* Immediate success of the procedure.
* Rate of patients with DAPT at < 1 month, 1-3 months, 3-6 months, and 6-12 months and relationship with the occurrence of events
* Composite endpoints:

Cardiac death, TV-MI and ID-TLR: (Target Lesion Failure (TLF)) Cardiac death, any myocardial infarction (MI) and ID-TVR: (Target Vessel Failure (TVF))

* Rate of overlapping devices: characteristics and relationship with occurrence of events
* Collection of imaging data of the cases where, according to the judgement of the investigator, intravascular imaging tests have been performed (IVUS, OCT).

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least 18 years of age at the time of signing the Informed Consent Form
* Patient is to be treated for de novo coronary lesions in a native coronary artery and amenable to receive a bioresorbable device
* The length of the treated lesion should be inferior to the nominal length of the device (12 mm, 18 mm, 28 mm) with a reference vessel diameter > 2 mm y < 3,8 mm.
* The patient will not have any relative contraindication for double antiplatelet therapy, with aspirin indefinitely and with a thienopyridine for at least 6 months

Exclusion Criteria:

* Cardiogenic shock
* Left main disease
* Aortocoronary graft
* Intrastent restenosis
* Potentially child-bearing women with no contraceptive methods
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with native coronary artery de novo lesions with indication for revascularization with a coronary device
Sampling Method: Non-Probability Sample
Enrollment: 2440 (Actual)
Dates: Start 2014-01; Primary Completion 2015-09 (Actual); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
MACE rate (major adverse cardiac events) at 12 months of follow-up: Cardiac death; Myocardial infarction; Target lesion revascularisation (TLR) ischemia-driven: Cardiac Death/All MI/ID-TLR | Clinical follow-up at 12 months

SECONDARY OUTCOMES:
Immediate success of the device/procedure | 1 day
Cardiac death | 12 months
Myocardial infarction | 12 months
Scaffold/Stent Thrombosis: Timing and Evidence | 12 months
Target lesion/vessel revascularization (TLR/TVR) | 12 months
Angina Events | 12 months
Rate of patients with DAPT at 12 months | 12 months
Rate of overlapping devices and characteristics | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Hernandez, MD, Principal Investigator — Seccion Hemodinamica y Cardiologia Intervencionista
Locations (1):
- Hospital 12 de Octubre, Madrid, Madrid, Spain